CLINICAL TRIAL: NCT00590616
Title: Utility of Clinical Examination in the Noninvasive Prediction of Aortic Atheroma - A Prospective Study
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 06-14035; 06-14035
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Atherosclerosis
Keywords: Aortic atheroma
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: transthoracic examination

INTERVENTIONS:
Procedure: transthoracic examination — observational transthoracic examination

SUMMARY:
Aortic atheroma has been correlated with traditional cardiac risk factors, coronary, carotid, renal and peripheral atherosclerosis, and is probably a manifestation of generalized atherosclerosis. Aortic atheroma has also been shown to be associated with atrial fibrillation, aortic valve sclerosis, and other calcification of the fibrous skeleton of the heart. None of the previous studies have looked at the noninvasive prediction of aortic atheroma using the history and physical signs of cardiovascular disease. This would be a time and cost-effective bedside diagnostic tool that would be useful prior to cardiac surgery, cardiac catheterization, and workup of ischemic stroke patients, especially when transesophageal echocardiogram (TEE) is being considered for diagnosis but cannot be obtained due to previously mentioned reasons. Although physical examination of peripheral vascular disease is non-specific, a combination of physical examination signs increases the probability of generalized atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who are referred for transesophageal echocardiography (TEE) since the primary endpoint is diagnosis of aortic atheroma on TEE

Exclusion Criteria:

* No exclusion after consent for TEE is obtained. Decision not to perform TEE at the discretion of treating physician

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for TEE examination, since the primary end-point would be diagnosis of aortic atheromatous disease on TEE. Prevalence of aortic atheroma, based on previous data at Creighton and other studies in any aortic atheroma ~50% and severe aortic atheroma ~5%.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2005-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Identify clinical predictors of aortic atheromatous disease and develop risk score to identify with reasonable accuracy the presence of any aortic atheromatous disease and severe atheromatous disease (grade 4 & 5). | 6 month. 1 year and 2 year

SECONDARY OUTCOMES:
Demonstrate the incremental value of physical exam signs to the history. | 6 month, 1 and 2 years
Follow-up on embolic events - transient ischemic attack (TIA), stroke and mortality and effect of medications | 6 months, 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Manu Kaushik, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States